CLINICAL TRIAL: NCT00408980
Title: is Dietary Manipulation of Human Milk Total Fat and Caloric Content Feasible?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: breastmilk.ctil
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2006-12-08 (Estimated); Status verified 2006-11

CONDITIONS: Breastfeeding
Keywords: diet; breast milk fat
MeSH Terms: conditions — Breast Feeding | interventions — CD36 Antigens; Caloric Restriction

INTERVENTIONS:
Behavioral: Fat and calorie controlled diet

SUMMARY:
The aim of this study is to verify whether dietary manipulations in lactating women allow increasing the fat and caloric content of human milk.

DETAILED DESCRIPTION:
The aim of this study is to verify whether dietary manipulations in lactating women allow increasing the fat and caloric content of human milk. specifically, we will test the following hypotheses:1) at constant caloric intake, 2 high fat (40% fat, 45% CHO) diets ( margarine e nriched versus butter enriched) lead to higher fat and caloric content of human milk than the low fat diet (5% fat, 80% CHO); and 2) All 3 groups will have strikingly different milk fatty acid profiles (mirroring the dietary fatty acid profile).

ELIGIBILITY:
Inclusion Criteria:

* breast feeding women
* healthy
* on no medications

Exclusion Criteria:

* women on medications

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Weinstadt Morya, MD, Principal Investigator — Shaare Zedek Medical Center, Jerusalem